CLINICAL TRIAL: NCT07340151
Title: Surgical Resection of Synchronous Pulmonary or Hepatic Oligometastatic Pancreatic Ductal Adenocarcinoma (PHOLIPANC) Following Pre-operative Liposomal Irinotecan Combined With Oxaliplatin and 5-Fluoracil/Folinic Acid (NALIRIFOX): A Phase II Open-Label Single Arm Trial
Brief Title: Resection/Synchronous Pulmonary or Hepatic Oligometastatic Pancreatic Ductal Adenocarcinoma
Acronym: PHOLIPANC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CTMS# 25-0006
Record Dates: First submitted 2025-12-22; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Adenocarcinoma of the Pancreas
Keywords: Oligometastatic disease; Hepatic oligometastatic adenocarcinoma of the pancreas; Pulmonary oligometastatic adenocarcinoma of the pancreas; Surgical resection

STUDY DESIGN:
Intervention Model Description: Interventional, open-label, non-randomized, single-arm clinical trial with 2 cohorts of participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Oligometastatic Cohort (Active Comparator): Participants who have pulmonary oligometastatic pancreatic tumor
  Interventions: Procedure: Surgical resection
- Liver Oligometastatic Cohort (Active Comparator): Participants who have hepatic oligometastatic pancreatic tumor
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — Patients with a technically resectable primary tumor and tumor response or stable disease of their metastatic disease according to the evaluation of an interdisciplinary tumor board after the first 4 cycles will undergo exploratory laparotomy and synchronous or staged resection of the primary tumor and the hepatic or pulmonary metastases by using the standard of care surgical techniques 2-6 weeks after the last neoadjuvant chemotherapy. Residual tumor classification, also known as R Classification defines how complete the resection of the malignancy has been at surgery: R0: no residual tumor/R1: microscopic residual tumor
  Other Names: R0/R1 resection

SUMMARY:
This is a clinical trial that tests a surgical treatment. Everyone in the study will get the same treatment, and there is no comparison or placebo group.

Patients can join the study if they have pancreatic cancer that has spread to only a few spots in the liver or lungs. They must be receiving a type of chemotherapy called NALIRIFOX before surgery (this is called neoadjuvant chemotherapy).

If the cancer gets worse during or after the first 4 cycles of chemotherapy, the patient will be removed from the study.

If the cancer stays the same or gets smaller after the first 4 cycles, doctors will check if the main tumor can be removed with surgery. If the tumor cannot be removed, the patient will get 4 more cycles of chemotherapy as standard of care.

If the main tumor can be removed, the patient will have surgery 2-6 weeks after finishing chemotherapy. During surgery, doctors will try to remove both the main tumor and the small tumors in the liver or lungs. If, during surgery, the doctor finds that the main tumor actually cannot be removed, the patient may receive 4 more cycles of chemotherapy starting 2-4 weeks after surgery.

DETAILED DESCRIPTION:
This is an interventional, open-label, non-randomized, single-arm clinical trial with 2 cohorts. Patients who have hepatic or pulmonary oligometastatic adenocarcinoma of the pancreas and who receive neoadjuvant Liposomal Irinotecan Combined with Oxaliplatin and 5-Fluoracil/Folinic Acid (NALIRIFOX) chemotherapy pre-operatively are eligible. In patients with progressive disease during or after the first four cycles, patients will become ineligible. Patients with tumor response or stable disease after the first 4 cycles but a non-resectable primary tumor according to the evaluation of an interdisciplinary tumor board will receive 4 more cycles of neoadjuvant chemotherapy as per standard of care. Patients with a technically resectable primary tumor and tumor response or stable disease of their metastatic disease according to the evaluation of an interdisciplinary tumor board after the first 4 cycles will undergo exploratory laparotomy and synchronous or staged resection of the primary tumor and the hepatic or pulmonary metastases by using the standard of care surgical techniques 2-6 weeks after the last neoadjuvant chemotherapy. If the primary tumor is deemed unresectable by the surgeon during exploratory laparotomy, these patients may receive 4 more cycles of adjuvant chemotherapy as per standard of care 2-4 weeks after the exploratory laparotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of treatment-naïve limited hepatic or pulmonary metastatic adenocarcinoma of the pancreas
2. Meet the definition of limited hepatic or pulmonary metastasis according to Computed Tomography/Magnetic Resonance Imaging (CT/MRI) that is done prior to the starting of any anticancer treatment. Either CT scan of chest, abdomen, and pelvis with intravenous contrast or a combination of MRI of abdomen and pelvis and CT scan of chest is acceptable radiographic imaging. CT/MRI can be done at an outside facility but must be reviewed by a local radiologist.

   * Definition of limited hepatic metastasis: 1 to 5 metastases in CT/MRI, which are potentially resectable or treatable by ablative procedures.

     * Note 1: Patients also fulfil this inclusion criterion if a hepatic metastasis was partly or entirely removed as part of the diagnosis and is thus not detectable by CT/MRI scan at screening.
     * Note 2: If more than 5 metastases are unexpectedly detected during surgery, it is not a violation of this inclusion criterion if the excess metastases had not been detectable by CT/MRI scan at screening.
   * Definition of limited pulmonary metastasis: 1 to 4 pulmonary nodules seen on CT/MRI, suspicious for pulmonary metastases as per the multidisciplinary tumor board radiologist and surgeon.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
4. Patients ≥18 years at the time of signing the informed consent
5. Being a candidate for chemotherapy with NALIRIFOX
6. Patient's written informed consent prior to any trial-specific procedure
7. Patient's legal capacity to consent to participation in the clinical trial.

Exclusion Criteria:

1. Acinar cell carcinoma and/or neuroendocrine carcinoma of the pancreas
2. Symptomatic clinically significant ascites
3. Evidence of any distant metastases other than limited hepatic or pulmonary metastasis as defined in inclusion criterion 1.
4. Evidence of simultaneous pulmonary and hepatic metastases
5. Any tumor-specific pretreatment of the adenocarcinoma of the pancreas (including but not limited to surgery, radiation therapy, chemotherapy or ablative procedures). Currently being on NALIRIFOX or its modified form is allowed, unless more than 2 treatments of NALIRIFOX have been given.
6. Any malignancies other than adenocarcinoma of the pancreas in the 2 years before the start of the clinical trial except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, breast cancer, prostate cancer or superficial bladder tumors (Ta, Tis and T1 staging where Ta=non-invasive; Tis=high-grade, flat non-invasive cancer in situ; T1=relatively small primary tumor that has not spread to surrounding tissues)
7. Known Human immunodeficiency virus (HIV) seropositivity
8. Known active or chronic Hepatitis B or Hepatitis C infection
9. Known glucuronidation deficiency (Gilbert's syndrome)
10. Any other severe concomitant disease or disorder, which could influence patient's ability to participate in the clinical trial and his/her safety during the trial or interfere with interpretation of results, e.g., severe hepatic, renal, pulmonary, cardiovascular, metabolic or psychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of R0/R1 resection | Prior to surgery to 4-12 weeks after surgery
  Assessed by tumor imaging

SECONDARY OUTCOMES:
Safety of surgical resection of synchronous pulmonary or hepatic oligometastatic ductal adenocarcinoma | End of surgical procedure
  Surgical complications will be defined based on Clavien-Dindo classification and will be monitored continuously. The monitoring rule will focus on Grade IIIa surgical complication or above deemed related to the chemotherapy regimen (liposomal irinotecan, oxaliplatin, 6-fluorouracil/folinic acid) which is beyond what may be expected for chemotherapy or resection without immunotherapy.
European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-30) | Prior to surgery and 4-12 weeks after surgery
  The QLQ-C30 is composed of both multi-item scales and single-item measures including 5 functional scales, 3 symptom scales, a global health status / QoL scale, and six single items.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  A crucial Summary Score (0-100) combines 13 scales (excluding Global QoL & Financial Impact), with higher scores indicating better overall quality of life. Scoring requires specific formulas from the official manual, with procedures for handling missing data and ensuring consistency across different scales, often involving reversing symptom scales for uniform interpretation.
European Organization for Research and Treatment of Cancer Quality of Life for pancreatic ductal adenocarcinoma (EORTC QLQ-PAN26) | Prior to surgery and 4-12 weeks after surgery
  Raw scores from the questionnaire items (e.g., 1=Not at all, 4=Very much) are linearly transformed to a 0-100 scale.
  Higher score on a symptom scale = Worse symptoms/more problems (e.g., pancreatic pain).
  Higher score on a functional scale = Better quality of life/functioning (e.g., planning activities)
Progression-free survival (PFS) | Up to 25 months after re-section of tumor
  Assessment of mortality of participant continuously post surgery until study end.
Recurrence-free survival (RFS) | Up to 25 months after re-section of tumor
  Assessment of health status of participant continuously post surgery until study end.
Overall survival | Up to 25 months after re-section of tumor
  Length of time participant survives post surgical re-section.

OTHER OUTCOMES:
Time to development of new/recurrent metastases | Up to 25 months after re-section of tumor
  Time to diagnosis of any new metastases or recurrence of resected tumor

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zheng, MD, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio